CLINICAL TRIAL: NCT06283771
Title: The Effect of Warmed Socks Developed as Wearable Technology on Hypothermia, Thermal Comfort Perception and Shivering in Healthy Volunteers
Brief Title: The Effect of Warmed Socks Developed as Wearable Technology on Hypothermia, Thermal Comfort Perception and Shivering
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Research Assistant, Tarsus University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: TU-BOZKUL-007
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Wearable Technology; Hypothermia; Shivering; Thermal Comfort Perception
MeSH Terms: conditions — Hypothermia | interventions — Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: The research was planned as a prospective, two-arm (1:1), randomized controlled, double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: An independent biostatistician, who is not involved in the study, will select 70 individuals from the list of students enrolled between 1-250 by computer-generated randomization. The information that the volunteers included in the research sample were assigned to group A (experimental) and B (control) according to the randomization table will be kept by the researcher and the socks with the same appearance, with and without heating feature will be numbered from 1 to 70 according to the randomization table and given to the researcher. Thus, the practitioner will be blinded as he/she does not know which sock has a heating feature and which one does not. Healthy volunteers will be blinded because they do not know which group they are in. The data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will also be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): The study group will wear heated socks to be developed with wearable technology
  Interventions: Other: Heated socks to be developed with wearable technology
- CONTROL GROUP (No Intervention): The control group will wear socks that look exactly the same as the heated socks developed with wearable technology worn by the study group, but with a closed heating circuit.

INTERVENTIONS:
Other: Heated socks to be developed with wearable technology — The study group will wear heated socks to be developed with wearable technology
  Arms: EXPERIMENTAL GROUP

SUMMARY:
In this study, it is aimed to reveal the effect of the use of heated socks to be developed as wearable technology by providing temperature control on body temperature, comfort perception level and shivering development in healthy volunteers and this purpose constitutes the unique value of the project. The research was planned as a prospective, two-arm (1:1), randomized controlled, double-blind study. The population of the study will consist of 4th year nursing students consisting of an average of 250 people who will enroll in the fall semester of the 2024-2025 academic year. As a result of the power analysis performed in the G*Power program, the sample will consist of 70 healthy volunteers, at least 35 in each group. In the study, data will be collected with the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form (Shivering Level Diagnosis Form and Temperature Comfort Perception Scale)" which includes the descriptive information of healthy volunteers. Healthy volunteers will fill out the "Introductory Characteristics Form" and "Hypothermia Monitoring Form" before being taken to the Faculty of Nursing Skills Laboratory for the application. Before the volunteers are taken to the single rooms in the laboratory, the environment will be cooled for 30 minutes with the air conditioner in the room so that the temperature is 21oC. The study group will wear socks developed with wearable technology and the control group will wear socks with the same appearance. The healthy volunteer will be asked to lie motionless on the bed for 60 minutes in a single room. Body temperature (with Braun tympanic thermometer), shivering level and temperature comfort perception will be recorded on the "Hypothermia Monitoring Form" when all healthy volunteers are taken to the Skills Laboratory, at 15 minutes, 30 minutes and 60 minutes, and when they leave the laboratory. The research data will be analyzed in a computer environment. Descriptive variables of healthy volunteers included in the study will be expressed as mean±standard deviation and median (maximum minimum), percentage and frequency. Changes in body temperature measurements obtained after wearing socks to be developed with wearable technology, repeated measurements, analysis of variance (Repeated ANOVA) if parametric, Friedman test if non-parametric, and post-hoc test will be used in intra-group multiple comparison analysis as further analy

DETAILED DESCRIPTION:
Increasing developments in science have led to rapid advances in health technology. One of these developments is wearable technology. Wearable devices play a key role in the field of healthcare, especially since they play an active role in providing data by monitoring changes in vital signs in real time. Textile-based sensors, electrodes and other devices are used in conjunction with wearable technological devices due to their low cost, flexibility and ease of application. Existing studies have focused on the impact of wearable technologies on positive patient outcomes in different fields. However, previously developed textile-based medical products, patents or utility model examples have not been designed to prevent hypothermia in healthy adults by providing temperature control. In this study, it is aimed to reveal the effect of the use of heated socks to be developed as wearable technology by providing temperature control on body temperature, comfort perception level and shivering development in healthy volunteers and this purpose constitutes the unique value of the project. The research was planned as a prospective, two-arm (1:1), randomized controlled, double-blind study. The population of the study will consist of 4th year nursing students consisting of an average of 250 people who will enroll in the fall semester of the 2024-2025 academic year. As a result of the power analysis performed in the G*Power program, the sample will consist of 70 healthy volunteers, at least 35 in each group, taking into account the losses with 95% power and a maximum of 5% type error in both directions. In the study, data will be collected with the "Descriptive Characteristics Form" and "Hypothermia Monitoring Form (Shivering Level Diagnosis Form and Temperature Comfort Perception Scale)" which includes the descriptive information of healthy volunteers. Healthy volunteers will fill out the "Introductory Characteristics Form" and "Hypothermia Monitoring Form" before being taken to the Faculty of Nursing Skills Laboratory for the application. Before the volunteers are taken to the single rooms in the laboratory, the environment will be cooled for 30 minutes with the air conditioner in the room so that the temperature is 21oC. The study group will wear socks developed with wearable technology and the control group will wear socks with the same appearance. The healthy volunteer will be asked to lie motionless on the bed for 60 minutes in a single room. Body temperature (with Braun tympanic thermometer), shivering level and temperature comfort perception will be recorded on the "Hypothermia Monitoring Form" when all healthy volunteers are taken to the Skills Laboratory, at 15 minutes, 30 minutes and 60 minutes, and when they leave the laboratory. The research data will be analyzed in a computer environment. Descriptive variables of healthy volunteers included in the study will be expressed as mean±standard deviation and median (maximum minimum), percentage and frequency. Changes in body temperature measurements obtained after wearing socks to be developed with wearable technology, repeated measurements, analysis of variance (Repeated ANOVA) if parametric, Friedman test if non-parametric, and post-hoc test will be used in intra-group multiple comparison analysis as further analysis.

ELIGIBILITY:
Inclusion Criteria:

* -Written and verbal permission to participate in the study was obtained,
* No communication problems,
* Speaks and understands Turkish,
* Non-hypothermic,
* Not diagnosed with a chronic disease,
* Not allergic to sock material,
* No peripheral vascular disease,
* Without a device that sends electric current into the body (pacemaker, etc.),
* Healthy volunteers with a body mass index within normal limits (18.5-24.9 kg/m2).

Exclusion Criteria:

* Written and verbal permission to participate in the research could not be obtained,
* Communication problems,
* Speaking Turkish but not understanding it,
* Diagnosed with a chronic disease,
* Hypothermic,
* Peripheral vascular disease,
* Allergic to sock material,
* A person with a device (pacemaker, etc.) that sends electric current into the body,
* Healthy volunteers with a body mass index not within normal limits (<18.5 kg/m2- >25 kg/m2)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Body temperature | 5 months
  Hypothermia Monitoring Form: It is a form in which body temperature, shivering level and temperature comfort perception of healthy volunteers are recorded. The body temperature of the healthy volunteers in the study and control groups will be measured when they are admitted to the basic skills laboratory, 15 minutes after they are admitted to the laboratory, 30 minutes after they are admitted to the laboratory, 60 minutes after they are admitted to the laboratory and when they leave the laboratory, and their shivering level and temperature comfort perception will also be measured during these periods. In this form, the measurement times of body temperature values were determined based on the literature
Shivering level | 5 months
  Tremor Level Diagnosis Form: The form, which Badjaita et al. (2008) determined the criteria by observation, determines the level of tremor according to the tremor in the extremities between 0 (no tremor) and 3 (severe tremor in the trunk, lower and upper extremities) points.
Thermal comfort perception | 5 months
  Hypothermia Monitoring Form: It is a form in which body temperature, shivering level and temperature comfort perception of healthy volunteers are recorded. The body temperature of the healthy volunteers in the study and control groups will be measured when they are admitted to the basic skills laboratory, 15 minutes after they are admitted to the laboratory, 30 minutes after they are admitted to the laboratory, 60 minutes after they are admitted to the laboratory and when they leave the laboratory, and their shivering level and temperature comfort perception will also be measured during these periods. In this form, the measurement times of body temperature values were determined based on the literature
Descriptive Characteristics | 5 months
  Descriptive Characteristics Form: The form created by the researcher in line with the literature consists of questions about descriptive characteristics of the voluntueers

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Bozkul, Principal Investigator — Tarsus University; Evren Değirmenci, Principal Investigator — Mersin University; Murat BOZLU, Principal Investigator — Mersin University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal DK, Viers BR, Rivera ME, Nienow DA, Frank I, Tollefson MK, Gettman MT. Physical activity monitors can be successfully implemented to assess perioperative activity in urologic surgery. Mhealth. 2018 Sep 26;4:43. doi: 10.21037/mhealth.2018.09.05. eCollection 2018. PMID 30363722
- [Background] Badjatia N, Strongilis E, Gordon E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Ostapkovich ND, Mayer SA. Metabolic impact of shivering during therapeutic temperature modulation: the Bedside Shivering Assessment Scale. Stroke. 2008 Dec;39(12):3242-7. doi: 10.1161/STROKEAHA.108.523654. Epub 2008 Oct 16. PMID 18927450
- [Background] Baskan, A., & Goncu-Berk, G. (2022). User Experience of Wearable Technologies: A Comparative Analysis of Textile-Based and Accessory-Based Wearable Products. Applied Sciences. 12(21), 11154. https://doi.org/10.3390/app122111154.
- [Background] Bayoumy K, Gaber M, Elshafeey A, Mhaimeed O, Dineen EH, Marvel FA, Martin SS, Muse ED, Turakhia MP, Tarakji KG, Elshazly MB. Smart wearable devices in cardiovascular care: where we are and how to move forward. Nat Rev Cardiol. 2021 Aug;18(8):581-599. doi: 10.1038/s41569-021-00522-7. Epub 2021 Mar 4. PMID 33664502
- [Background] Burns A, Adeli H. Wearable technology for patients with brain and spinal cord injuries. Rev Neurosci. 2017 Nov 27;28(8):913-920. doi: 10.1515/revneuro-2017-0035. PMID 28850551
- [Background] Castellani JW, Young AJ. Human physiological responses to cold exposure: Acute responses and acclimatization to prolonged exposure. Auton Neurosci. 2016 Apr;196:63-74. doi: 10.1016/j.autneu.2016.02.009. Epub 2016 Feb 21. PMID 26924539